CLINICAL TRIAL: NCT07332793
Title: Mechanisms of Precise Immune Cell Phenotyping and Prognostic Prediction in Severe Infection
Acronym: PIC-PSI
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2025-03-137
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Sepsis
Keywords: immune cells; Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples collected during routine clinical care, retained for immune cell analysis and related laboratory assessments. No samples will be used for DNA extraction or genetic analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Infection ICU Cohort: Adult patients with severe infection admitted to the intensive care unit (ICU). All participants receive standard clinical care as determined by their treating physicians. No experimental interventions are assigned.

SUMMARY:
The goal of this observational study is to learn how changes in immune cells are linked to outcomes in adults with severe infection who are treated in the intensive care unit (ICU). Severe infections, including sepsis, can affect how the immune system works and may lead to poor recovery or death. Researchers want to better understand these immune changes so that people at higher risk can be identified earlier.

The main questions this study aims to answer are:

Are certain immune cell patterns linked to survival or death within 28 days? Are these immune patterns linked to organ failure or longer stays in the ICU? Participants will be adults with severe infection who are admitted to the ICU as part of their routine medical care. This study does not change or add to their medical treatment.

Participants will:

Have small blood samples collected at several time points during their ICU stay Allow researchers to review their medical records, including test results and outcomes Researchers will analyze immune cells in the blood and relate these findings to clinical outcomes. The results may help improve future risk assessment and understanding of immune changes in people with severe infection.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study conducted in adult patients with severe infection who are admitted to the intensive care unit (ICU). The study aims to characterize dynamic changes in immune cell profiles during critical illness and to examine how these changes are associated with short-term clinical outcomes.

Severe infection, including sepsis, is frequently accompanied by profound alterations in immune function. While some individuals recover, others develop persistent organ dysfunction or die despite standard medical care. Current clinical and laboratory markers provide limited information about immune status and do not reliably predict outcomes. A more detailed understanding of immune cell patterns in critically ill patients may help improve risk stratification and future clinical decision-making.

Adult patients (aged 18 years or older) who are diagnosed with severe infection according to established clinical criteria and admitted to the ICU will be screened for eligibility. Participants will be enrolled consecutively after informed consent is obtained from the patient or a legally authorized representative. This study does not involve any experimental intervention, and all participants will receive standard medical care as determined by their treating clinicians.

Peripheral blood samples will be collected at predefined time points during the ICU stay, including early and later phases of illness. These samples will be used to assess immune cell populations and their activation states using established laboratory methods. In addition, routinely collected clinical data will be recorded, including demographic information, severity of illness scores, laboratory test results, organ support measures, and clinical outcomes.

The primary clinical outcome of interest is all-cause mortality within 28 days after ICU admission. Secondary outcomes include the development of organ dysfunction and length of ICU stay. Immune cell data will be analyzed in relation to these outcomes to identify immune patterns that are associated with different clinical trajectories.

Statistical analyses will focus on describing immune cell distributions, identifying immune phenotypes using data-driven approaches, and evaluating associations between immune patterns and clinical outcomes while accounting for relevant clinical variables. The results of this study are intended to improve understanding of immune alterations in severe infection and to inform future research aimed at improving prognosis assessment and patient management.

All data will be collected and stored in accordance with ethical and regulatory requirements. Participant confidentiality will be maintained through coded identifiers, and access to identifiable information will be restricted to authorized study personnel.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Admission to the intensive care unit (ICU)
* Diagnosis of severe infection, including sepsis, based on established clinical criteria
* Enrollment within the early phase of ICU admission
* Informed consent obtained from the patient or a legally authorized representative

Exclusion Criteria:

* Age younger than 18 years
* Pregnancy or breastfeeding
* Known history of hematologic malignancy or active solid malignancy receiving chemotherapy
* Known primary immunodeficiency or long-term immunosuppressive therapy prior to ICU admission
* Human immunodeficiency virus (HIV) infection with severe immunosuppression
* Previous enrollment in this study
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years or older who are admitted to the intensive care unit (ICU) with severe infection, including sepsis. Participants are enrolled during the early phase of ICU admission and receive standard clinical care as determined by their treating physicians. This observational study does not involve assignment to experimental interventions.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-01-16 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | Within 28 days after ICU admission
  All-cause mortality assessed within 28 days after admission to the intensive care unit.

SECONDARY OUTCOMES:
ICU length of stay | Length of stay in the intensive care unit, measured in days from ICU admission to ICU discharge.
  From ICU admission to ICU discharge
Organ dysfunction | Organ dysfunction assessed using routinely collected clinical data during the first 28 days after ICU admission.
  Within 28 days after ICU admission
Secondary infection | Within 28 days after ICU admission
  Secondary infection during ICU stay
GPCR Expression on Regulatory T Cells | At baseline (ICU admission), Day 7, and Day 14
  The expression levels of selected G protein-coupled receptors (GPCRs) on peripheral blood regulatory T cells (Tregs), quantified by flow cytometry and expressed as mean fluorescence intensity (MFI) and/or percentage of positive cells.
Molecular phenotypes of immune cells | At ICU admission and during ICU stay
  Molecular phenotypes of peripheral immune cell subsets, will be assessed by multiparameter flow cytometry.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive clinical information, and data sharing is not covered by the current ethics approval. Data will be used solely for the purposes specified in the approved study protocol.